CLINICAL TRIAL: NCT02958280
Title: A Tailored Physical Activity Smartphone App for Patients With Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1604-003; R33AA024295 (NIH)
Record Dates: First submitted 2016-09-27; First posted 2016-11-08 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Dependence
Keywords: Exercise; Smartphone
MeSH Terms: conditions — Alcoholism; Motor Activity | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Advice Plus the Fit&Sober App (Experimental): Phase 1 (app development & Open Pilot) will consist of: 1) development of the Fit&Sober prototype; 2) series of usability studies with patients with AUDs; and 3) An open pilot of a 12-week trial (n=20) to test the feasibility and acceptability of the Fit&Sober app with patients with AUDs in early recovery.
  Phase 2: RCT of the Fit&Sober app with 160 patients with AUD
  Interventions: Behavioral: Fit&Sober App; Behavioral: Brief Advice
- Brief Advice for Physical Activity (Active Comparator): Phase 2: Participants randomized to the BA only condition will meet for a 30-minute discussion with a research staff member. In this session, participants will receive information about the public health guidelines for physical activity, the benefits of physical activity for physical and mental health, as well as sobriety, strategies for getting started as well as instruction on gradually increasing physical activity
  Interventions: Behavioral: Brief Advice

INTERVENTIONS:
Behavioral: Fit&Sober App — Fit&Sober is a smartphone-based physical activity app that includes multilevel strategies for increasing physical activity for patients with AUDs in early recovery.
  Arms: Brief Advice Plus the Fit&Sober App
Behavioral: Brief Advice — Participants randomized to the BA only condition will meet for a 30-minute discussion with a research staff member. In this session, participants will receive information about the public health guidelines for physical activity, the benefits of physical activity for physical and mental health, as well as sobriety, strategies for getting started as well as instruction on gradually increasing physical activity

SUMMARY:
The purpose of the study twofold: first, a smartphone-based physical activity application (app), which will be called Fit&Sober, will be developed and tailored specifically for patients with alcohol use disorders (AUDs); then, the feasibility, acceptability, and short-term increases in physical activity with the use of the Fit&Sober app will be examined over the course of a 12-week intervention.

DETAILED DESCRIPTION:
Alcohol Use Disorders (AUDs) are highly prevalent and a costly public health problem. AUDs are the third leading preventable cause of death in the U.S. and are associated with significant negative physical and psychological health consequences, costing the U.S. economy an estimated $235 billion dollars per year. While progress has occurred in developing treatments for AUDs, relapse rates are still extremely high, ranging from 60-95% in first year following treatment. Given the compelling evidence for the benefits of increased physical activity for physical health, psychological functioning, and drinking outcomes, efforts to help patients with AUDs adopt and sustain increased levels of physical activity (PA) are likely to result in significant public health impact. Capitalizing on the advantages for scalability and dissemination afforded by the use of technology, the investigators will develop a smartphone-based physical activity application (app), which will be called Fit&Sober, tailored specifically for patients with AUDs. Although a number of PA apps exist, the majority suffer from a lack of theory-based concepts known to influence behavior change. Grounded in Self Determination Theory (SDT) and Social Cognitive Theory (SCT), the investigators will develop and tailor the Fit&Sober app for patients with AUDs by designing features that will help patients develop intrinsic, value-driven goals (e.g., exercising for benefits related to sobriety) with a focus on increasing the saliency of immediate rewards associated with PA (e.g., decreased alcohol urges and improved affect). The investigators propose that why someone exercises makes a difference for long-term PA. Early recovery from AUDs, when negative affect is a risk for relapse and urges to drink are common, may be an opportune time to help patients develop internalized, self-determined motivation through experientially making connections between exercise and acute improvements in affect and cravings. Smartphone technology offers unique advantages for self-monitoring these changes in affect and cravings in relation to physical activity. The aims of the proposed study include:

Phase 1: App Development and Open Pilot

1. A Mixed-methods approach will be used to develop a tailored, theoretically-driven smartphone intervention (Fit&Sober App) to help patients in early recovery from AUDs increase levels of physical activity.

1. a. The principles of agile software development will be used to create a prototype of the app. Feedback obtained through a series of usability studies and focus groups with patients with AUDs will iteratively inform subsequent versions of the app.
2. To conduct an open pilot trial with 20 patients with AUDs in early recovery to determine the feasibility, acceptability, and short-term increases in PA with use of the Fit&Sober app. After 12-weeks of app use:

2.a. Through self-report measures and qualitative interviews, feedback will be obtained on use of the Fit&Sober app as well satisfaction with the app, strengths and weaknesses of the app, any challenges encountered with the app, suggestions for areas of improvement, and adverse events.

2.b. Through examination of the Fit&Sober metadata, indicators of the extent of app usage (e.g., days utilized, time spent on the application, components accessed, etc.) will be obtained.

2.c. Through objectively measured PA, short-term increases in physical activity levels will be examined.

Phase 2 -- RCT Aims

1. To conduct a preliminary, randomized controlled trial of the Fit&Sober App compared to Brief Advice (BA) for Exercise among 160 patients in early recovery from AUDs. We hypothesize that, compared to BA, Fit&Sober will be associated with:

   1. Higher levels of short-term (3-month) and long-term (6-,12-month), objective-measured moderate-to-vigorous physical activity and sedentary behaviors
   2. Higher percent days abstinent (PDA) from alcohol and lower levels of depression and anxiety symptoms at each follow-up
   3. Higher levels of theoretically-relevant, PA-related mediating variables including: self-efficacy, positive outcome expectancies, and self-determined motivation at 3- and 6-month follow-ups
2. To explore the relationship between usage of app features and levels of physical activity engagement

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age,
* meet DSM-5 criteria for alcohol use disorder as assessed by the SCID-P,
* are sedentary, (i.e., less than 60 minutes of moderate-intensity exercise per week for the past 6 months), and
* are currently engaged in alcohol treatment.

Exclusion Criteria:

* current DSM-5 diagnosis moderate/severe substance use disorder or anorexia or bulimia nervosa
* a history of psychotic disorder or current psychotic symptoms
* current suicidality or homicidality,
* current mania
* marked organic impairment according to either the medical record or responses to the diagnostic assessments,
* physical or medical problems that would not allow safe participation in a program of moderate intensity physical activity (i.e., not medically cleared by study physician),
* current pregnancy or intent to become pregnant during the next 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate-to-vigorous physical activity per week | 12-months
  Measured by accelerometry

SECONDARY OUTCOMES:
Satisfaction with App | 12 Weeks
  System Usability Scale
App Usage | 12 weeks
  metadata collected from app
Alcohol Abstinence | 12-months
  Percent days abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abrantes AM, Meshesha LZ, E Blevins C, Battle CL, Lindsay C, Marsh E, Feltus S, Buman M, Agu E, Stein M. A Smartphone Physical Activity App for Patients in Alcohol Treatment: Single-Arm Feasibility Trial. JMIR Form Res. 2022 Oct 19;6(10):e35926. doi: 10.2196/35926. PMID 36260381